CLINICAL TRIAL: NCT03944057
Title: An Open-Label, Single-Arm Study of ATG-010 Plus Dexamethasone in Patients With Multiple Myeloma Refractory to Prior Treatment With Immunomodulatory Agents and Proteasome Inhibitor
Brief Title: A Study of Evaluating the Safety and Efficacy of ATG-010 in Relapsed Refractory Multiple Myeloma
Acronym: MARCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-MM-001
Record Dates: First submitted 2019-04-30; First posted 2019-05-09 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Relapse/Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — selinexor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ATG-010 + Dexamethasone (Experimental): Open-label ATG-010 80mg plus Dexamethasone 20 mg
  Interventions: Drug: ATG-010

INTERVENTIONS:
Drug: ATG-010 — ATG-010 (Selinexor) will be given at an oral fixed milligram (mg) dose of 80 mg twice weekly each week for four-week cycles (total of 8 ATG-010 doses per cycle).
  Dexamethasone 20 mg will be given with each dose of ATG-010 (Selinexor)
  Other Names: Selinexor

SUMMARY:
This is an open-label, single-arm study of ATG-010 (selinexor) plus low-dose Dexamethasone (Sd) in patients with multiple myeloma previously treated with lenalidomide and bortezomib refractory to prior treatment with immunomodulatory agents and proteasome Inhibitors.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter study of ATG-010 (Selinexor) plus low dose Dexamethasone dosed twice weekly each week in four-week cycles, in patients with triple-refractory MM. The population refractory for the primary efficacy analysis will contain only patients with triple-MM enrolled. PK analysis would be performed which would contain approximately 30% of the patients enrolled. Safety analyses will be performed on the overall population of patients who received at least one dose of study drug among triple-refractory patient populations. Patients will receive treatment until progressive disease (PD), death, toxicity that cannot be managed by standard care, or withdrawal, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with federal, local, and institutional guidelines.
2. Age ≥ 18 years at the time of signing informed consent.
3. Patients must have previously received including proteasome inhibitors (PI) (i.e., lenalidomide) and immunomodulatory drugs (i.e., bortezomib) and were refractory to both drugs.
4. Any clinically significant non-hematological toxicities (except for peripheral neuropathy as described in exclusion criterion #17) that patients experienced from treatments in previous clinical studies must have resolved to Grade ≤ 2 by Cycle 1 Day 1.
5. Adequate hepatic function within 21 days prior to Cycle 1 Day 1: total bilirubin < 2x upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3x ULN), AST < 2.5x ULN and ALT < 2.5x ULN.
6. Adequate renal function within 21 days prior to Cycle 1 Day 1: estimated creatinine clearance of ≥ 20 mL/min, calculated using the formula of cockroft and gault.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
8. Measurable MM based on IMWG guidelines.
9. Adequate hematopoietic function within 21 days prior to Cycle 1 Day 1 (See Exclusion Criterion #20 for transfusion washout periods for RBCs and platelets):

   1. Hemoglobin level ≥ 8.5 g/dL
   2. ANC ≥ 1000/mm^3
   3. Platelet count ≥ 75,000/mm^3 (patients in whom < 50% of bone marrow nucleated cells are plasma cells) or ≥ 50,000/mm^3 (patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells. [Platelet transfusions < 1 week prior to Cycle 1 Day 1 are prohibited (see below).]
10. Female subjects of child-bearing potential must have both of the following:

    1. Agree to the use of two study physician-approved contraceptive methods simultaneously, or practice complete abstinence starting at the time of ICF signature, while on study medication, and 3 months following the last dose of study drug.
    2. Have negative serum pregnancy test result at screening.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Active smoldering MM.
  2. Active plasma cell leukemia.
  3. Documented systemic amyloid light chain amyloidosis.
  4. Active central nervous system (CNS) MM.
  5. Pregnancy or breastfeeding.
  6. Chemotherapy ≤ 4 week, radiation and immunotherapy ≤ 4 weeks prior to Cycle 1 Day 1, and radio-immunotherapy 6 weeks prior to Cycle 1 Day 1.
  7. Active graft vs. host disease (after allogeneic stem cell transplantation) at Cycle 1 Day 1
  8. Life expectancy of < 4 months.
  9. Major surgery within four weeks prior to Cycle 1 Day 1.
  10. Active, unstable cardiovascular function:

      1. Symptomatic ischemia, or
      2. Uncontrolled clinically-significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics are excluded; patients with 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block/right bundle branch block (LAFB/RBBB) will not be excluded), or
      3. Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥ 3, or
      4. Myocardial infarction (MI) within 3 months prior to Cycle 1 Day 1.
  11. Prior exposure to a SINE compound, including ATG-010.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jiao, MD, Study Director — Medical Monitor
Locations (17):
- China (17):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guanzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central Suoth University, Changsha, Hunan
  - The First Affilate Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital Affiliate Shanghai JiaoTong University, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - Tianjin blood research institute, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Qiu L, Xia Z, Fu C, Chen W, Chang C, Fang B, An G, Wei Y, Cai Z, Gao S, Weng J, Chen L, Jing H, Li F, Liu Z, Chen X, Liu J, Wang A, Yu Y, Xiang W, Lynch K, Yu Z, Fu W. Selinexor plus low-dose dexamethasone in Chinese patients with relapsed/refractory multiple myeloma previously treated with an immunomodulatory agent and a proteasome inhibitor (MARCH): a phase II, single-arm study. BMC Med. 2022 Apr 5;20(1):108. doi: 10.1186/s12916-022-02305-4. PMID 35379237

RESULTS

PARTICIPANT FLOW:
Groups:
- ATG-010 + Dexamethasone: Open-label ATG-010 80mg plus Dexamethasone 20 mg
  ATG-010: ATG-010 (Selinexor) will be given at an oral fixed milligram (mg) dose of 80 mg twice weekly each week for four-week cycles (total of 8 ATG-010 doses per cycle).
  Dexamethasone 20 mg will be given with each dose of ATG-010 (Selinexor)
Period: Overall Study
Arm/Group | ATG-010 + Dexamethasone
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ATG-010 + Dexamethasone
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 82
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23 (3.29)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The primary efficacy endpoint of ORR consists of proportion of patients who achieve PR, VGPR, CR, or sCR according to IMWG 2016 criteria:
  * CR means Negative IFE of serum and urine, disappearance of any soft tissue plasmacytomas (SPD), and <5% plasma cells in bone marrow aspirates;
  * sCR means CR as defined above plus normal FLC ratio and absence of clonal cells in bone marrow biopsy by immunohistochemistry (κ/λ ratio ≤ 4:1 or ≥ 1:2 for κ and λ patients, respectively, after counting ≥ 100 plasma cells);
  * VGPR means Serum and urine M-protein detectable by IFE but not on electrophoresis, or ≥90% reduction in serum M-protein plus urine M-protein level <100 mg per 24 hours;
  * PR means ≥50% reduction of serum M-protein plus reduction in 24-hour urine M-protein by ≥90% or to <200 mg per 24 hours. If the serum and urine M-protein are unmeasurable, a ≥50% decrease in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ATG-010 + Dexamethasone
Number analyzed (Participants) | 82
Participants | 24

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: To evaluate progression-free survival
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | ATG-010 + Dexamethasone
Number analyzed (Participants) | 82
month | 3.7 [2.02 to 4.66]

ADVERSE EVENTS:
Time Frame: From study drug dosed to 30 days after last study drug dose. SAE was collected from consent. The period is at least no less than 12 months.
Arm/Group | ATG-010 + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 7/82
Serious Adverse Events (participants affected / at risk) | 45/82
Other Adverse Events (participants affected / at risk) | 82/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATG-010 + Dexamethasone (N=82)
Peumonia (Infections and infestations) | 12
Platelet count dicreased (Investigations) | 12
Upper respiratory infection (Infections and infestations) | 4
Anemia (Blood and lymphatic system disorders) | 4
White blood cell count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATG-010 + Dexamethasone (N=82)
Decreased platelet count (Investigations) | 72
Decreased white-cell count (Investigations) | 68
Lymphocyte count decreased (Investigations) | 63
Neutrophil count decreased (Investigations) | 59
Weight loss (Investigations) | 54
Aspartate aminotransferase increased (Investigations) | 20
Alanine aminotransferase increased (Investigations) | 19
Blood lactate dehydrogenase increased (Investigations) | 16
γ-glutamyltransferase increased (Investigations) | 15
Serum creatinine increased (Investigations) | 11
C-reactive protein increased (Investigations) | 10
Total protein decreased (Investigations) | 9
Blood Urea increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 8
Amylase Increased (Investigations) | 6
Lipase increased (Investigations) | 6
β2-microglobulin increased (Investigations) | 6
α-hydroxybutyrate dehydrogenase increased (Investigations) | 5
Glucose increased (Investigations) | 5
Hyponatremia (Metabolism and nutrition disorders) | 56
Decreased appetite (Metabolism and nutrition disorders) | 51
Hyperglycemia (Metabolism and nutrition disorders) | 47
Hypocalcemia (Metabolism and nutrition disorders) | 36
Hypokalaemia (Metabolism and nutrition disorders) | 31
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26
Hypophosphatemia (Metabolism and nutrition disorders) | 19
Hyperuricemia (Metabolism and nutrition disorders) | 16
Hypertriglyceridemia (Metabolism and nutrition disorders) | 13
Hypochloridemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypoproteinemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 5
Nausea (Gastrointestinal disorders) | 64
Vomiting (Gastrointestinal disorders) | 42
Diarrhea (Gastrointestinal disorders) | 25
Constipation (Gastrointestinal disorders) | 14
Month ulcer (Gastrointestinal disorders) | 7
Anemia (Blood and lymphatic system disorders) | 71
Adynamia (General disorders) | 49
Fatigue (General disorders) | 13
Oedema peripheral (General disorders) | 9
Fever (General disorders) | 8
Lung infection (Infections and infestations) | 25
Infection upper respiratory (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 5
Dizzy (Nervous system disorders) | 15
Hypaesthesia (Nervous system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Sleeplessness (Psychiatric disorders) | 18
Tachycardia sinus (Cardiac disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 7
Vision blurred (Eye disorders) | 10
Cataracts (Eye disorders) | 5
Hypertension (Vascular disorders) | 6
Pruritis (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT03944057/Prot_SAP_000.pdf